CLINICAL TRIAL: NCT04168814
Title: An Observational Study of the Nutritional Status in Locally Advanced or Metastatic Solid Cancer Patients While Receiving Immunotherapy in Spain: the NutriOncoSearch (NOS) Study
Brief Title: Nutritional Status in Locally Advanced or Metastatic Solid Cancer Patients in Spain: the NutriOncoSearch (NOS) Study
Acronym: NOS
Status: Completed | Type: Observational
Sponsor: Universidad Pontificia Comillas (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Iqvia Pty Ltd (Industry); SPANISH SOCIETY OF ONCOLOGY NURSING (Unknown)
Responsible Party: Principal Investigator, Julio C. de la Torre-Montero, Principal Investigator, professor, Universidad Pontificia Comillas
Other Study IDs: SEEO-19-01-NOS
Record Dates: First submitted 2019-11-14; First posted 2019-11-19 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Malnutrition; Oncologic Complications; Oncology; Quality of Life
Keywords: Nutritional status; Oncology Patients; Anticancer treatments; Quality of Life
MeSH Terms: conditions — Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oncology patients (Immunotherapy alone or in combination)): 1. Outpatients, over 18 years old, with locally advanced or metastatic solid tumors (with the idea of homogenizing the sample as far as possible and in line with what has been published up to now, also stratified in line with Globocan).
  2. Patients under targeted active treatment either exclusively or in combination with chemotherapy or radiotherapy. Targeted therapy (immunotherapy) defined with: PD1, PDL1 inhibitors. At least 12 weeks of treatment.
  Interventions: Other: Observational test
- Oncology Patients (Chemo-Radiotherapy group).: 1. Outpatients, over 18 years old, with locally advanced or metastatic solid tumors (with the idea of homogenizing the sample as far as possible and in line with what has been published up to now, also stratified in line with Globocan).
  2. Patients under active treatment either in combination with chemotherapy or radiotherapy. At least 12 weeks of treatment.
  Interventions: Other: Observational test

INTERVENTIONS:
Other: Observational test — Nutritional risk (NutriScore), based on weight, weight loss, tumor location, and treatment, Nutritional status (VGS, Global Subjective Assessment Valoración Global Subjetiva, in Spanish), ECOG performance status; nutritional therapy (oral nutritional supplements, enteral nutrition, parenteral nutrition, dietary advice); type of treatment: chemo, type of chemo, adjuvant, neoadjuvant, palliative, curative endocrine therapy, targeted therapy +-immunotherapy vs QQT/RT therapy; cancer site. Covid-19 diagnosis.

SUMMARY:
Malnutrition is a common medical problem in oncology patients. It is well known that the presence of malnutrition negatively affects patients' evolution and their quality of life, increasing the incidence of infection, hospital stay, and mortality.

The new knowledge of cancer biology has made it possible to know the mechanisms of cancer progression.

New treatments have been developed thanks to this knowledge including molecular target treatments aimed at these cancer mechanics and to reverse the antitumor capacity of the immune system. However, these treatments have different toxicities than classic and anachronistic treatments such as chemotherapy and radiotherapy, including alterations in glucose metabolism, endocrinopathies, rhabdomyolysis, etc. that can alter both the patient's nutritional status and quality of life. Additionally, a deficient nutritional status can have an impact on the intestinal microbiota, compromising the efficacy of the new antitumor treatments.

The principal objective of this study is to characterize the nutritional status of the cancer outpatient receiving immunotherapy through a screening performed in Hospital consultations in Spain.

Secondary Endpoints are (a). To describe the percentage of patients that receive nutritional counseling or nutritional support (enteral and/or parenteral nutrition) among those diagnosed as malnourished or at risk. And (b) to categorize the percentage and descriptive characteristics of cancer patients with mild, moderate, or severe malnutrition that goes to a hospital consultation in Spain and describe the percentage and descriptive characteristics of patients with malnutrition according to sociodemographic and clinical characteristics.

DETAILED DESCRIPTION:
Study Title:

An observational study of the Nutritional status in locally advanced or metastatic solid cancer patients while receiving immunotherapy in Spain: the NutriOncoSearch (NOS) study.

Research Question:

What is the current nutritional status in advanced cancer patients receiving immunotherapy or any other targeted therapies in Spain?

Study Background & Rationale:

Malnutrition is a common medical problem in oncology patients. Between 15 and 40% of patients with cancer present weight loss at diagnosis and the incidence of malnutrition increases over the course of the disease until 80% of all cancer patients. It is well known that the presence of malnutrition negatively affects patients' evolution and their quality of life, increasing the incidence of infection, hospital stay, and mortality.

The new knowledge of cancer biology has made it possible to know the mechanisms of cancer progression. These mechanisms include:

1. Self-sufficiency in growth signals.
2. Insensitivity to anti-growth signals.
3. Evading apoptosis.
4. No breaks in the replicate potential
5. Sustained angiogenesis. New treatments have been developed thanks to this knowledge including molecular target treatments aimed at these cancer mechanics and to reverse the anti-tumor capacity of the immune system. However, these treatments have different toxicities than classic and anachronistic treatments such as chemotherapy and radiotherapy, including alterations in glucose metabolism, endocrinopathies, rhabdomyolysis, etc. that can alter both the patient's nutritional status and quality of life. Additionally, a deficient nutritional status can have an impact on the intestinal microbiota, compromising the efficacy of the new anti-tumor treatments.

Regarding the nutritional status of cancer patients, some studies have been developed. In France, a 1-day prospective prevalence survey was carried out in 154 public or private hospital wards in 24 French cities. The investigators were to include all patients with cancer who were present at the hospital on the day of the survey and who agreed to participate. The results of this study showed a high prevalence of malnutrition (39%) and a high rate of malnourished patients not receiving nutrition support (42.4%). Recently, the PreMio study (Italy) assessed the nutritional status of cancer patients on their first visit for care. Findings showed that first-visit PreMiO patients were often malnourished or at risk for malnutrition when they entered the study- 40% to 80% of patients had signs and indicators of nutritional impairment- even in early disease stages, particularly in gastroesophageal, pancreatic, head and neck, and colorectal cancer patients.

In Spain, two old studies analyzed the nutritional situation of Spanish oncology patients. The first one is a multicentric study published in 2005 with data from outpatients and hospitalized patients. In this study, the scored PG-SGA indicated that 52% of the patients were moderately or severely malnourished and, of the total population analyzed, 97.6% required some form of nutritional recommendation to prevent, or reverse malnutrition. Since then, only the sub-analysis of the PREDYCES study gave information on the nutritional status of cancer patients (hospitalized) in our country (8). This analysis revealed that 36.4% of hospitalized oncology patients were at nutritional risk at the time of hospital discharge. It also demonstrated its significant association with longer hospital stays and higher healthcare costs. Despite all of this, only 1/3 of patients at nutritional risk received nutritional support. There are little data on the nutritional status of non-hospitalized oncology patients and, to our knowledge, none of them analyzed the effects of new target therapies. As these new therapies represent the future of oncology, it´s of most importance to understand what this effect is. The aim of this observational study is to determine the prevalence of malnutrition (or risk of malnutrition) in the Spanish population of outpatients that receive immunotherapy or any other targeted therapies For that end the investigators would like to explore nutritional status using validated tools like NutriScore, and Global Subjective assessment, Spanish version.

Study Design

Study Type: Clinical Non-Interventional

Condition to be studied and incidence: Nutritional status

Due to the epidemiologic characteristics of this study, the investigators don´t ask about adverse events or their relationship with specific drugs: the investigators will ask for generic groups of agents or treatments.

Study Population (ages, gender, relevant disease states): Adult patients, both sexes, Stages III-IV all solid cancers.

Duration of subject participation: This a descriptive, prospective and analytic study. Patients will be asked once, and no more.

The total number of subjects to be enrolled: 610 subjects.

* The number of study or comparison groups: two 2:1 relation. 408 patients with immunotherapy with or without chemotherapy or radiotherapy and 204 with chemotherapy or radiotherapy alone, both of them in the first line of treatment,
* The study will be performed on multiple different days: the recruitment will be concomitant and limited to a minimum of 30 and a maximum of 70 patients depending on the number of patients the center deals with. The estimation is that each center will dedicate from one to two weeks to recruit the total number of patients.

Specific details of Treatment/Intervention: (prescription and/or therapy, devices, equipment, solutions, product to be used in conducting the study:

Not applicable.

Efficacy Assessments Not applicable.

Statistical Methods (for analyzing primary & secondary endpoints):

Descriptive statistics like clinical and sociodemographic characteristics of the studied population will be expressed by means and SDs for the continuous variables and frequency distribution for the qualitative variables. The investigators will use the ӽ2 test and Fisher exact test for the qualitative data set and Student t-test for quantitative data, with a significance level of .05 and a confidence interval of 95%. Multivariate logistic regression analysis and odds ratios can be efficiently conducted as a measure of statistical correlation to link nutrition status and associated factors.

Based on the number of cancer diagnoses in 2019 in Spain (REDECAN), there will be an incidence of 277.234 new cases, with a prevalence of 772.853 cases (5-years projection). With this population the investigators calculate a proportion estimation, with a confidence interval 1-α of 99%, d= 3%, p= 0,5, the sample size is 504, with an expected loss of (R=)15% sample size is 610 subjects. Investigators propose a stratification in two groups, in a 2:1 proportion, 408 patients in the immunotherapy-only group and 204 patients in the control, chemotherapy-in-combination group.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients, over 18 years old, with locally advanced or metastatic solid tumors (with the idea of homogenizing the sample as far as possible and in line with what has been published up to now, also stratified in line with Globocan).
2. Patients under immunotherapy treatment either exclusively or in combination with chemotherapy or radiotherapy. Immunotherapy defined by checkpoint treatments inhibitors PD-1, PDL-1 y CTLA-4. At least 12 weeks of treatment.

Key Exclusion Criteria:

1. Estimated survival below 12 weeks (palliative criteria).
2. Patients that meet diagnostic criteria (DSM-IV and ICD-10) of nervous anorexia and bulimia.
3. Patients with severe psychiatric disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total number of subjects to be enrolled: 610 subjects, counting lost.
  * Number of study or comparison groups: two.
  * The study will be performed on multiple different days: the recruitment will be concomitant and limited to a minimum of 30 patients depending on the number of patients the center deals with. The estimation is that each center will dedicate from an estimation of twelve weeks to recruit the total number of patients.
Sampling Method: Non-Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Six months
  To characterize the nutritional status of the cancer outpatient receiving either immunotherapies or any other targeted therapies through a screening performed in Hospital consultations in Spain.

SECONDARY OUTCOMES:
Nutritional counselling | Six months
  To describe the percentage of patients that receive nutritional counselling or nutritional support (enteral and/or parenteral nutrition) among those diagnosed as malnourished or at risk.
Descriptive characteristic mild, moderate or severe malnutrition | Six months
  To categorize the percentage and descriptive characteristic of cancer patients with mild, moderate or severe malnutrition that goes to a hospital consultation in Spain and describe the percentage and descriptive characteristic of patients with malnutrition according to sociodemographic and clinical characteristics (type of tumor and TNM stage).

CONTACTS AND LOCATIONS:
Overall Officials: Julio C de la Torre-Montero, Ph.D, Principal Investigator — Comillas Pontifical University
Locations (11):
- Spain (11):
  - Hospital Virgen de los Lirios, Alcoy, Alicante
  - Hospital Universitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Universidad Pontificia Comillas, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Universitario Donosti, San Sebastián
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Dissemination in biomedical research journals
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting March 2021
Access Criteria: Open Access

REFERENCES:
- [Background] de Las Penas R, Majem M, Perez-Altozano J, Virizuela JA, Cancer E, Diz P, Donnay O, Hurtado A, Jimenez-Fonseca P, Ocon MJ. SEOM clinical guidelines on nutrition in cancer patients (2018). Clin Transl Oncol. 2019 Jan;21(1):87-93. doi: 10.1007/s12094-018-02009-3. Epub 2019 Jan 8. PMID 30617923
- [Background] Arribas L, Hurtos L, Sendros MJ, Peiro I, Salleras N, Fort E, Sanchez-Migallon JM. NUTRISCORE: A new nutritional screening tool for oncological outpatients. Nutrition. 2017 Jan;33:297-303. doi: 10.1016/j.nut.2016.07.015. Epub 2016 Aug 13. PMID 27751743
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Escortell Sanchez R, Reig Garcia-Galbis M. [ENTERAL NUTRITION ON THE NUTRITIONAL STATUS OF CANCER]. Nutr Hosp. 2015 Oct 1;32(4):1408-16. doi: 10.3305/nh.2015.32.4.9227. Spanish. PMID 26545500
- [Background] Gomez-Candela C, Luengo LM, Cos AI, Martinez-Roque V, Iglesias C, Zamora P, Gonzalez-Baron R. [Subjective global assessment in neoplastic patients]. Nutr Hosp. 2003 Nov-Dec;18(6):353-7. Spanish. PMID 14682183
- [Result] Hebuterne X, Lemarie E, Michallet M, de Montreuil CB, Schneider SM, Goldwasser F. Prevalence of malnutrition and current use of nutrition support in patients with cancer. JPEN J Parenter Enteral Nutr. 2014 Feb;38(2):196-204. doi: 10.1177/0148607113502674. PMID 24748626
- [Result] Segura A, Pardo J, Jara C, Zugazabeitia L, Carulla J, de Las Penas R, Garcia-Cabrera E, Luz Azuara M, Casado J, Gomez-Candela C. An epidemiological evaluation of the prevalence of malnutrition in Spanish patients with locally advanced or metastatic cancer. Clin Nutr. 2005 Oct;24(5):801-14. doi: 10.1016/j.clnu.2005.05.001. PMID 15993517
- [Result] Muscaritoli M, Lucia S, Farcomeni A, Lorusso V, Saracino V, Barone C, Plastino F, Gori S, Magarotto R, Carteni G, Chiurazzi B, Pavese I, Marchetti L, Zagonel V, Bergo E, Tonini G, Imperatori M, Iacono C, Maiorana L, Pinto C, Rubino D, Cavanna L, Di Cicilia R, Gamucci T, Quadrini S, Palazzo S, Minardi S, Merlano M, Colucci G, Marchetti P; PreMiO Study Group. Prevalence of malnutrition in patients at first medical oncology visit: the PreMiO study. Oncotarget. 2017 Aug 10;8(45):79884-79896. doi: 10.18632/oncotarget.20168. eCollection 2017 Oct 3. PMID 29108370
- [Result] Planas M, Alvarez-Hernandez J, Leon-Sanz M, Celaya-Perez S, Araujo K, Garcia de Lorenzo A; PREDyCES(R) researchers. Prevalence of hospital malnutrition in cancer patients: a sub-analysis of the PREDyCES(R) study. Support Care Cancer. 2016 Jan;24(1):429-435. doi: 10.1007/s00520-015-2813-7. Epub 2015 Jun 23. PMID 26099900
- See also: SEOM, Las cifras del cáncer en España. Cancer database in Spain, year 2019. — https://seom.org/dmcancer/wp-content/uploads/2019/Informe-SEOM-cifras-cancer-2019.pdf